CLINICAL TRIAL: NCT00450866
Title: Phase II Trial of Patupilone in Patients With Brain Metastases From Breast Cancer
Brief Title: Epothilone B in Treating Patients With CNS Metastases From Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David Peereboom, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, David Peereboom, MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE5106; P30CA043703 (NIH); MSKCC-07036 (Other: MSKCC)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2013-10-09 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Breast Cancer; Metastatic Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; tumors metastatic to brain; leptomeningeal metastases; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Brain Neoplasms; Meningeal Carcinomatosis; Breast Neoplasms, Male | interventions — epothilone B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Epothilone B (Experimental)
  Interventions: Biological: epothilone B

INTERVENTIONS:
Biological: epothilone B — Patupilone will be administered as a single intravenous infusion over 20 minutes, once every 3 weeks. Patupilone will be administered at a dose of 10 mg/m2 (q3weeks) with actual body weight.
  Other Names: Patupilone

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as epothilone B, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well epothilone B works in treating patients with CNS metastases from breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 3-month CNS-progression free survival of patients with CNS metastases secondary to breast cancer treated with epothilone B.

Secondary

* Determine the toxicity of this drug in these patients.
* Determine the CNS response rate and duration of CNS response in patients treated with this drug.
* Determine the systemic disease response rate and duration of systemic response in patients treated with this drug.
* Determine the overall survival of patients treated with this drug.

OUTLINE: This is a multicenter, open-label study.

Patients receive epothilone B IV over 20 minutes on day 1. Courses repeat every 21 days in the absence of disease progression, satisfactory response, or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed carcinoma of the breast
* CNS metastases (i.e., brain parenchymal lesions and/or leptomeningeal disease), meeting 1 of the following criteria:

  * Recurrent or progressive CNS metastases after whole brain radiotherapy

    * If only evaluable site of CNS progression has been previously treated with stereotactic radiosurgery, radiation necrosis must be excluded by radiographic (e.g., positron emission tomography scan or magnetic resonance spectroscopy) or histologic assessment
  * Newly diagnosed, untreated, asymptomatic brain or leptomeningeal metastases
* Patient must be neurologically stable, as demonstrated by a stable dose of steroids and anticonvulsants for ≥ 1 week prior to obtaining baseline gadolinium-enhanced MRI of the brain and/or ≥ 1 week prior to beginning study treatment
* No CNS complications requiring urgent neurosurgical intervention (e.g., resection or shunt placement)
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* Karnofsky performance status 60-100%
* Life expectancy ≥ 3 months
* Absolute neutrophil count > 1,500/mm^3
* Hemoglobin > 9.0 g/dL
* Platelet count > 100,000/mm^3 (red blood cell transfusion and repeat evaluation allowed)
* Bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT < 2.5 times ULN
* Alkaline phosphatase < 2.5 times ULN
* Creatinine < 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* No known hypersensitivity to epothilones
* No peripheral neuropathy > grade 1
* No unresolved diarrhea within the past 7 days

  * Grade 0 diarrhea required at study entry
* No concurrent serious medical illness (e.g., HIV positivity or active hepatitis B or C)
* No severe cardiac insufficiency (e.g., New York Heart Association class III-IV heart disease) with uncontrolled and/or unstable cardiac or coronary artery disease
* No active or suspected acute or chronic uncontrolled infection, including abscess or fistulae
* No other malignancy within the past 3 years except curatively treated nonmelanoma skin cancer, prostate cancer, or carcinoma in situ of the cervix
* No history of noncompliance to medical regimens or inability or unwillingness to return for all scheduled visits
* No contraindications to MRI, including any of the following:

  * Pacemaker
  * Ferromagnetic implants
  * Claustrophobia
  * Extreme obesity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 2 weeks since prior noncytotoxic drugs (e.g., small molecule-targeted drugs) and recovered
* More than 3 weeks since prior cytotoxic chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* More than 3 weeks since prior intracranial surgery and recovered
* More than 4 weeks since prior radiotherapy and recovered
* More than 4 weeks since prior major surgery
* More than 28 days since prior investigational compounds or drugs
* No prior epothilones
* No concurrent known diarrheagenic agents
* No other concurrent anticancer agents, including investigational agents, biological agents, or chemotherapy
* No other concurrent experimental therapies
* Concurrent hormone therapy and/or trastuzumab (Herceptin®) allowed
* No concurrent Coumadin® or other agents containing warfarin

  * Low dose Coumadin® (≤ 1 mg) for prophylactic maintenance of indwelling lines or ports allowed
* No concurrent radiotherapy for central metastases (e.g., vertebral or mediastinal metastases)

  * Concurrent radiotherapy for local peripheral metastases not being used as marker lesions allowed
* No concurrent prophylactic hematopoietic growth factors during course 1
* No concurrent herbal or nontraditional medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-01; Primary Completion 2011-06 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Peereboom, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center; Joseph Baar, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter conducted at the Cleveland Clinic, University Hospitals Case Medical Center, Massachusetts General Hospital, Memorial Sloan Kettering Cancer Center, and the University of Michigan.Fifty five patients were treated on this study between February 2007 and May 2010, all of whom are considered eligible.
Groups:
- Epothilone B (Group A): Group A: Patients with progressive, radiographically measurable parenchymal brain metastases after whole brain radiation therapy (WBRT). Patupilone will be administered as a single intravenous infusion over 20 minutes, once every 3 weeks. Patupilone will be administered at a dose of 10 mg/m2 (q3weeks) with actual body weight.
- Epothilone B (Group B): Group B: an exploratory cohort of patients, with either leptomeningeal metastases (LMD) or unirradiated, asymptomatic brain metastasis from breast cancer (BCBM).Patupilone will be administered as a single intravenous infusion over 20 minutes, once every 3 weeks. Patupilone will be administered at a dose of 10 mg/m2 (q3weeks) with actual body weight.
Period: Overall Study
Arm/Group | Epothilone B (Group A) | Epothilone B (Group B)
Started | 45 | 10
Completed | 38 | 7
Not Completed | 7 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Death | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Epothilone B (Groups A and B): Epothilone B : Patupilone will be administered as a single intravenous infusion over 20 minutes, once every 3 weeks. Patupilone will be administered at a dose of 10 mg/m2 (q3weeks) with actual body weight.
Arm/Group | Epothilone B (Groups A and B)
Number analyzed (Participants) | 55
Age, Continuous [Median (Full Range); unit: years] | 50 (8.6) [31 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 48
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 55
Central Nervous System (CNS) metastases [Number; unit: participants] — Group A: Patients with progressive, radiographically measurable parenchymal brain metastases after whole brain radiation therapy (WBRT) Group B: an exploratory cohort of patients, with either leptomeningeal metastases (LMD) or unirradiated, asymptomatic brain metastasis from breast cancer (BCBM).
  participants
    Group A | 45
    Group B | 10

OUTCOME MEASURES:

1. Primary Outcome: Central Nervous System (CNS) Progression-free Survival(PFS)
Description: The number of patients that are documented to have progression free survival at 3 months after treatment. Progression free is define as <25% increase in tumor area.
  PFS will be measured from the date of entry into the trial to the date of documented progression of brain metastases or death.
Time Frame: 3 months after treatment
Population: Intention to treat
Measure: Number; unit: participants
Groups:
- Epothilone B: Group A: Group A: Patients with progressive, radiographically measurable parenchymal brain metastases after whole brain radiation therapy (WBRT). Patupilone will be administered as a single intravenous infusion over 20 minutes, once every 3 weeks. Patupilone will be administered at a dose of 10 mg/m2 (q3weeks) with actual body weight.
- Epothilone B: Group B: Group B: an exploratory cohort of patients, with either leptomeningeal metastases (LMD) or unirradiated, asymptomatic brain metastasis from breast cancer (BCBM).Patupilone will be administered as a single intravenous infusion over 20 minutes, once every 3 weeks. Patupilone will be administered at a dose of 10 mg/m2 (q3weeks) with actual body weight.
Arm/Group | Epothilone B: Group A | Epothilone B: Group B
Number analyzed (Participants) | 45 | 10
participants | 12 | 2

2. Secondary Outcome: Toxicity as Measured by NCI CTCAE v3.0
Description: Percent of patients that experience the most common grade 3 and above toxicities possibly related to study drug - to be measured using the NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 3.0.
Time Frame: 3 months after treatment
Population: Intention to treat
Measure: Number; unit: percentage of participants
Arm/Group | Epothilone B (Groups A and B)
Number analyzed (Participants) | 55
percentage of participants | 44

3. Secondary Outcome: CNS Response Rate, for Measurable Disease Will be Assessed by the Modified McDonald Criteria
Description: Complete Response (CR): the circumstance when the tumor is no longer seen by neuroimaging Partial Response (PR): Decrease of >50% in the product of two diameters Stable Disease (SD): the circumstance when the scan shows no change. Progression (P): a > 25% increase in tumor area (two diameters)
Time Frame: 3 months after treatment
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Epothilone B: Group A | Epothilone B: Group B
Number analyzed (Participants) | 45 | 10
participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 5 | 0
  Stable Disease (SD) | 9 | 2
  Progression (P) | 31 | 8

4. Secondary Outcome: Systemic Disease Response Rate for Measurable Disease Will be Assessed by the Modified McDonald Criteria
Description: as for outcome 3
Time Frame: 3 months after treatment
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Epothilone B (Groups A and B)
Number analyzed (Participants) | 55
participants
  Complete Response (CR) | 1
  Partial Response (PR) | 7
  Stable Disease (SD) | 18
  Progression (P) | 29

5. Secondary Outcome: Overall Survival
Description: Median time (months) that patients survived during the duration of the study.
Time Frame: 48 months from start of study
Population: Intention to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Epothilone B (Groups A and B)
Number analyzed (Participants) | 55
months | 12.7 [6.6 to 21]

ADVERSE EVENTS:
Time Frame: Adverse events were collected while patients were on study over a 4 year period.
Arm/Group | Epothilone B (Groups A and B)
Serious Adverse Events (participants affected / at risk) | 18/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epothilone B (Groups A and B) (N=55)
Anemia (Blood and lymphatic system disorders) | 1
Aphasia (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Death not associated with CTCAE term - Death NOS (not otherwise specified) (General disorders) | 1
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 1
Dehydration (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 8
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) Total (General disorders) | 1
Hemorrhage, upper GI (Gastrointestinal disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pain - Abdomen NOS (not otherwise specified) (Gastrointestinal disorders) | 1
Pain - Head/headache (Nervous system disorders) | 1
Pain, thorax (related to persistent coughing) (Respiratory, thoracic and mediastinal disorders) | 1
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1
Renal Insufficiency (Renal and urinary disorders) | 1
Syncope (fainting) (Nervous system disorders) | 1
Ulcer, GI - Duodenum (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Weakness hand, left (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epothilone B (Groups A and B) (N=55)
Abdominal Pain (Gastrointestinal disorders) | 15
Alopecia (Skin and subcutaneous tissue disorders) | 9
Anemia (Blood and lymphatic system disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 20
Ataxia (Nervous system disorders) | 4
Constipation (Gastrointestinal disorders) | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dehydration (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 45
Dizziness (Nervous system disorders) | 11
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 4
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 11
Edema: limb (Vascular disorders) | 5
Fatigue (asthenia, lethargy, malaise) (General disorders) | 48
Flatulence (Gastrointestinal disorders) | 3
Heartburn/dyspepsia (Gastrointestinal disorders) | 8
Hypokalemia (Investigations) | 6
Insomnia (General disorders) | 3
Memory impairment (Nervous system disorders) | 3
Mood alteration - Anxiety (Psychiatric disorders) | 5
Mood alteration - Depression (Psychiatric disorders) | 3
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 7
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 6
Nausea (Gastrointestinal disorders) | 32
Neuropathy: sensory (Nervous system disorders) | 18
Neutropenia (Blood and lymphatic system disorders) | 4
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 12
Pain - Head/headache (Nervous system disorders) | 18
Pain-Back (Musculoskeletal and connective tissue disorders) | 4
Pain-Bone (Musculoskeletal and connective tissue disorders) | 5
Pain-Joint (Musculoskeletal and connective tissue disorders) | 7
Pain-Muscle (Musculoskeletal and connective tissue disorders) | 8
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6
Sore throat (Gastrointestinal disorders) | 3
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 5
Visual Changes (Eye disorders) | 6
Vomiting (Gastrointestinal disorders) | 20
Weight loss (Investigations) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes